CLINICAL TRIAL: NCT06611839
Title: A Multicenter, Single-Arm Phase I/II Clinical Study of the Venetoclax, Ivosidenib, and Azacitidine Triple-Drug Regimen in the Treatment of Chemotherapy-eligible Adult Patients With IDH1-Mutated Acute Myeloid Leukemia.
Brief Title: Venetoclax in Combination With Ivosidenib and Azacitidine for Newly Diagnosed IDH1-Mutated AML
Acronym: IDH1-AML-2024
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIT2024067
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: AML; IDH1 Mutation; Treatment
MeSH Terms: interventions — ivosidenib; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax、Ivosidenib and Azacitidine (Experimental): The study was divided into two phases: dose climbing (phase I)and dose extension (phase II).
  Interventions: Drug: Ivosidenib, Venetoclax, Azacitidine

INTERVENTIONS:
Drug: Ivosidenib, Venetoclax, Azacitidine — phase I: Induction therapy：Ivosidenib 、Venetoclax、Azacitidine
  Dose climbing stage: adopt the 3 + 3 design principle, and the dose level 0,-1and 1 are set as follows
  dose level 0: Ivosidenib 500mg d1-28 Venetoclax 100mg d-3，200mg d-2，400mg d-1,800mg d1-14 Azacitidine 75mg/m2/d, d1-7
  dose level -1:Ivosidenib 500mg d1-28 Venetoclax 100mg d-3，200mg d-2，400mg d-1, 600mg d1-14 Azacitidine 75mg/m2/d, d1-5
  dose level 1:Ivosidenib 500mg d1-28 Venetoclax 100mg d-3，200mg d-2，400mg d-1 800mg d1-21 Azacitidine 75mg/m2/d, d1-7
  Consolidation therapy intermediate-dose cytarabine regimen ： 3 courses
  If IDH1 mutant residual disease was positive before consolidation chemotherapy, Ivosidenib was added;
  Maintenance treatment:
  Azacitidine、Venetoclax 、Ivosidenib： 6 courses
  phase II: dose based on phase I results

SUMMARY:
Venetoclax can bind to the BCL-2 protein, thereby initiating the apoptosis program and exerting anti-AML effects. The induction regimen combining venetoclax with hypomethylating agents (HMA) significantly improves the remission rate (over 60%) in elderly unfit AML patients and markedly prolongs survival in those achieving complete remission. Isocitrate dehydrogenase (IDH) 1 and 2 are involved in the citric acid cycle. Approximately 20% of AML patients carry IDH1 or IDH2 mutations, which lead to the reduction of α-ketoglutarate to 2-hydroxyglutarate (2-HG). 2-HG can cause histone methylation and inhibit TET2 activity, resulting in DNA hypermethylation, thereby affecting gene expression and cell differentiation. IDH mutations are more common in elderly patients and are often associated with cytogenetic abnormalities; they may also co-occur with FLT3-ITD, NPM1, or DNMT3A mutations. Ivosidenib is an IDH1 inhibitor, and previous studies have confirmed its safety and efficacy in AML treatment. According to adult AML treatment guidelines, IDH-mutated patients eligible for intensive chemotherapy may receive IDH inhibitors during induction therapy. Based on the study by Montesinos et al. on the role of ivosidenib and azacitidine in IDH-mutated AML, for patients ineligible for intensive chemotherapy, a new treatment option has been added: IDH1-mutated AML patients may receive ivosidenib (500 mg, days 1-28) combined with azacitidine (75 mg/m²/day for 7 days) in 28-day cycles, or ivosidenib monotherapy. Recent studies have shown that a triple-drug regimen comprising ivosidenib, venetoclax, and azacitidine demonstrates excellent efficacy and safety. In chemotherapy-ineligible patients, the triple regimen achieved a composite complete remission rate (CRc) of 86% and an overall response rate (ORR) of 92%. At a median follow-up of 27.4 months, the 2-year overall survival (OS) was 72%, and the 2-year event-free survival (EFS) was 72%. Therefore, this study aims to conduct a multicenter, single-arm clinical trial to determine the maximum tolerated dose of the triple-drug regimen (ivosidenib, venetoclax, and azacitidine) and preliminarily evaluate the long-term efficacy of this combination. Additionally, it seeks to elucidate the relationship between measurable residual disease (MRD) levels and the selection of transplantation treatment strategies, providing evidence for MRD-based therapeutic decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet AML according to WHO (2022) or AML and MDS/AML defined by ICC standards with IDH1 mutations detected by PCR or second-generation sequencing.
2. Age ≥14 years old, male or female.
3. The physical status assessment (ECOG-PS) of the Eastern Oncology Collaboration group was 0-2 points.
4. Fulfill the requirements of the following laboratory tests (performed within 7 days prior to treatment) :

   1. Total bilirubin ≤ 1.5 times the upper limit of normal value (same age);
   2. AST and ALT≤ 2.5 times the upper limit of normal value (same age);
   3. Blood creatinine < 2 times the upper limit of normal (same age);
   4. Myocardial enzymes < 2 times the upper limit of normal (same age);
   5. Left ventricular ejection fraction >50% by measure of echocardiogram (ECHO) Informed consent must be signed before the commencement of all specific study procedures, and is signed by the patient himself or his immediate family. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the condition, the informed consent shall be signed by the legal guardian or the patient's immediate family.

Exclusion Criteria:

Subjects who meet any of the following criteria are excluded from the study:

1. Acute promyelocytic leukemia with PML-RARA fusion gene
2. Acute myeloid leukemia with RUNX1-RUNX1T1 or CBFB-MYH11 fusion gene
3. Acute myeloid leukemia with BCR-ABL fusion gene
4. Treated patients (but can receive hydroxyurea or cytarabine to lower tumor burden).
5. Concurrent malignant tumors of other organs (those requiring treatment).
6. Active heart disease, defined as one or more of the following:

   1. A history of uncontrolled or symptomatic angina;
   2. Myocardial infarction less than 6 months after enrollment;
   3. Have a history of arrhythmia requiring drug treatment or severe clinical symptoms;
   4. Uncontrolled or symptomatic congestive heart failure (> NYHA level 2);
7. Serious infectious diseases (uncured tuberculosis, pulmonary aspergillosis).
8. Those who were not considered suitable for inclusion by the researchers.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
CRc rate | Efficacy was assessed at least 2 weeks after completion of the first course of induction therapy.
  The ratio of patients achieved CR/CRh/CRi.
CRc MRD negtive rate by flow cytometry | Efficacy was assessed at least 2 weeks after completion of the first course of induction therapy.
  The CRc MRD negtive rate was detected by flow cytometry after induction, consolidation and maintenance therapy.
CRc MRD negtive rate by PCR | Efficacy was assessed at least 2 weeks after completion of the first course of induction therapy.
  The CRc MRD negtive rate was detected by PCR after induction, consolidation and maintenance therapy.
The maximum tolerated dose of ivosidenib and venetoclax combined with intensive chemotherapy | up to 3 months after enrollment of the first participants
  To determine the maximum tolerated dose of ivosidenib and venetoclax combined with intensive chemotherapy

SECONDARY OUTCOMES:
Event-free survival (EFS) | up to 2 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of failed to achieve complete remission, the date of relapse, or the date of death, whichever occurred first.
overall survival | up to 2 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of death or the date of last follow-up, whichever occurred first.
Relapse free survival | up to 2 years after the date of the last enrolled participants
  The interval from CR to the date of relapse, or the date of death, or the date of last follow-up, whichever occurred first.
30-day mortality | Within 30 days of the date of the last enrolled participants
  Percentage of patients who died within 30 days from enrollment
60-day mortality | Within 60 days of the date of the last enrolled participants
  Percentage of patients who died within 60 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, MD, Principal Investigator — Blood diseases hospital
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China